CLINICAL TRIAL: NCT03013530
Title: Assessment of Factors Involved in the Decision-making for ICU Patients' Care
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0296
Record Dates: First submitted 2016-12-19; First posted 2017-01-06 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Decision Making
Keywords: Intensive care unit; Triage and Therapy.; Advance Directives (AD).; Simulation model of real situations. (hypothetical scenario); Intensivist physician.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Patients with chronic disease
  Interventions: Procedure: Decision making for ICU patients' care

INTERVENTIONS:
Procedure: Decision making for ICU patients' care — Study of factors involved in the decision-making for ICU patients' care. Effect of advance directives (AD).

SUMMARY:
A new law about the advance directives (AD) has been recently voted in France on February 2, 2016. This " Claeys-Leonetti " law has made the AD more binding, as in other countries. This should lead to a greater respect of the human autonomy principle. However, the interpretation of these guidelines is often difficult and may differ between doctors. Indeed, the subjectivity of these interpretations could lead to different medical decisions by physicians.

The investigators intend to assess the effect of advance directives (AD) on decision making in care by intensivists, using a simulated (hypothetical) situation.

DETAILED DESCRIPTION:
Observational simulation (hypothetical) study of intensivist decisions for selected real patients.

Each patient writes advance directives (AD) after receiving clear information (videos and interview with an independent intensivist).

Intensivists answer to 5 questions for two simulations (hypothetical) models (scenario) on pneumonia and occlusive syndrome, in 3 times: without the AD, with AD, and with AD by knowing the drafting conditions (information from intensivist).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients :
* 20 patients with chronic diseases or 80 years old patient or older,
* 4 patients with chronic cardiac failure challenged in heart transplant
* 4 patients with chronic renal failure challenged in kidney transplant
* 4 COPD patients in terminal stage
* 4 patients with lung cancer challenged in surgery
* 4 patients, 80 years old or older, without cognitive impairment

Inclusion criteria for physician :

* Working in Intensive Care Unit (ICU)
* From the 10 ICUs involved in the protocol

Exclusion Criteria:

* Exclusion criteria for physician :
* Decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients' care
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Intensivists's answers to 5 questions for the 2 scenarios for each of the 20 patients | at day 1
  Intensivists's answers to 5 questions for the 2 scenarios for each of the 20 patients, in 3 times: without AD first, then with AD and AD with knowing they were made with an intensivist, in this order

SECONDARY OUTCOMES:
Comparison of answers to 5 questions for the 2 scenarios for each of the 20 patients between the 3 scenarios submission time for each intensivist (intra-individual variability). | at day 1
Comparison for each question | at day 1
Assessment of the concordance between the AD and the intensivists's answers. Direct comparison for objective criteria (organ replacement) between the patients's AD and intensivists's answers. And expert opinion for subjective criteria | at day 1
Drafting time for the realization of the AD | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre LAUTRETTE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Smirdec M, Jourdain M, Guastella V, Lambert C, Richard JC, Argaud L, Jaber S, Klouche K, Medard A, Reignier J, Rigaud JP, Doise JM, Chabanne R, Souweine B, Bourenne J, Delmas J, Bertrand PM, Verdier P, Quenot JP, Aubron C, Eisenmann N, Asfar P, Fratani A, Dellamonica J, Terzi N, Constantin JM, Van Lander A, Guerin R, Pereira B, Lautrette A. Impact of advance directives on the variability between intensivists in the decisions to forgo life-sustaining treatment. Crit Care. 2020 Dec 2;24(1):672. doi: 10.1186/s13054-020-03402-7. PMID 33267904